CLINICAL TRIAL: NCT04760977
Title: Prehospital Management of Hypotensive Trauma in HEMS
Acronym: SPITFIRE
Status: Recruiting | Type: Observational
Sponsor: Azienda Usl di Bologna (Other Government)
Responsible Party: Sponsor
Other Study IDs: 959-2020-OSS-AUSLBO
Record Dates: First submitted 2021-02-16; First posted 2021-02-18 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Hypotension and Shock; Wounds and Injuries; Emergencies; Critical Care
Keywords: Transportation of Patients; Wounds and Injuries; Emergencies; Critical Care
MeSH Terms: conditions — Hypotension; Shock; Wounds and Injuries; Emergencies | interventions — Administration, Inhalation; Blood Transfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trauma patients in shock: The study focuses on hypotensive trauma patients assisted by HEMS teams
  Interventions: Drug: Drugs administration; Device: Resuscitative endovascular balloon occlusion of the aorta; Biological: Blood transfusions; Other: Prehospital management; Device: Prehospital eFAST

INTERVENTIONS:
Drug: Drugs administration — Antifibrinolytics, analgesics, sedatives, neuromuscular blocking agents
Device: Resuscitative endovascular balloon occlusion of the aorta — Resuscitative technique for exsanguinating traumas
  Other Names: REBOA
Biological: Blood transfusions — Transfuion of transported blood products for exsanguinating traumas
Other: Prehospital management — Stay and play strategy vs scoop and run
Device: Prehospital eFAST — Prehospital thorax/abdomen extended focused assessment sonography for trauma

SUMMARY:
Up to today, inadequate evidences and knowledge exist about the best prehospital management of hypotensive trauma patients and its clinical consequence on the in-hospital recovery and mortality.

Also new emerging therapies such as prehospital blood transfusion and REBOA (resuscitative endovascular balloon occlusion of the aorta) are lacking strong evidences in, eventually, reducing hospital mortality and improving outcomes.

Moreover, prehospital emergency medicine is throughout Italy an heterogeneous system that has no unique standard operating procedures and, even among HEMS (helicopter emergency medical service), management and therapies on complex trauma patients may vary upon local policies.

With this study we aim to enroll hypotensive trauma patients and study factors of prehospital rescue that can be associated with in-hospital mortality and recovery, eventually even with hospital outcome. For each patients data as demographic, kind of trauma (mechanism, injury scores), therapies and maneuvers will be recorded and then analyzed in comparison with in-hospital data such as need for transfusion, ABG parameters, length of stay (in-ward and ICU), need of therapies like invasive ventilation and renal replacement therapy, recovery and outcome

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Witnessed traumatic event managed by HEMS
* Shock at first evaluation (Systolic blood pressure < 90 mmHg)
* Suspect or obvious ongoing haemorrage

Exclusion Criteria:

* Patients in cardiac arrest at HEMS arrival in which resuscitation is not started or interrupted by HEMS crew

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population object of study is represented by all the trauma patients managed by the HEMS crew that are experiencing a probable or obvious haemorragic shock
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
30 days mortality | 30 days

SECONDARY OUTCOMES:
survival from prehospital to hospital admmission | 1 day
Hospital length of stay | 6 months
Blood products transfused during the first 24 hours after hospital admission | 24 hours
Transport time | 24 hours
  time from dispatch to hospital admission (if any)

CONTACTS AND LOCATIONS:
Locations (16):
- Italy (16):
  - Ospedale di Alessandria, Alessandria
  - Base HEMS Aosta, Aosta
  - Ospedale di Bolzano, Bologna
  - Base HEMS Borgo Sesia, Borgosesia
  - Base HEMS Cuneo-Levaldigi, Cuneo
  - Ospedale Careggi Firenze, Florence
  - Ospedale di Siena, Ospedale di Pisa, Grosseto
  - Ospedale di Siena, Ospedale di Pisa, Massa
  - Ospedale di Padova, Padua
  - Pavullo HEMS base, Pavullo nel Frignano
  - Pieve di Cadore HEMS base, Pieve di Cadore
  - Ospedale di Torino, Torino
  - Base HEMS Trento, Trento
  - Treviso hospital, Treviso
  - Udine FVG, Udine
  - Ospedale di Verona Borgo Trento, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brown JB, Sperry JL, Fombona A, Billiar TR, Peitzman AB, Guyette FX. Pre-trauma center red blood cell transfusion is associated with improved early outcomes in air medical trauma patients. J Am Coll Surg. 2015 May;220(5):797-808. doi: 10.1016/j.jamcollsurg.2015.01.006. Epub 2015 Jan 24. PMID 25840537
- [Result] Smith IM, James RH, Dretzke J, Midwinter MJ. Prehospital Blood Product Resuscitation for Trauma: A Systematic Review. Shock. 2016 Jul;46(1):3-16. doi: 10.1097/SHK.0000000000000569. PMID 26825635
- [Result] Spahn DR, Bouillon B, Cerny V, Duranteau J, Filipescu D, Hunt BJ, Komadina R, Maegele M, Nardi G, Riddez L, Samama CM, Vincent JL, Rossaint R. The European guideline on management of major bleeding and coagulopathy following trauma: fifth edition. Crit Care. 2019 Mar 27;23(1):98. doi: 10.1186/s13054-019-2347-3. PMID 30917843
- [Result] Powell EK, Hinckley WR, Gottula A, Hart KW, Lindsell CJ, McMullan JT. Shorter times to packed red blood cell transfusion are associated with decreased risk of death in traumatically injured patients. J Trauma Acute Care Surg. 2016 Sep;81(3):458-62. doi: 10.1097/TA.0000000000001078. PMID 27050884
- [Result] Brohi K, Gruen RL, Holcomb JB. Why are bleeding trauma patients still dying? Intensive Care Med. 2019 May;45(5):709-711. doi: 10.1007/s00134-019-05560-x. Epub 2019 Feb 11. No abstract available. PMID 30741331
- [Derived] Tartaglione M, Carenzo L, Gamberini L, Lupi C, Giugni A, Mazzoli CA, Chiarini V, Cavagna S, Allegri D, Holcomb JB, Lockey D, Sbrana G, Gordini G, Coniglio C; SPITFIRE Study Collaborators. Multicentre observational study on practice of prehospital management of hypotensive trauma patients: the SPITFIRE study protocol. BMJ Open. 2022 May 30;12(5):e062097. doi: 10.1136/bmjopen-2022-062097. PMID 35636792